CLINICAL TRIAL: NCT06174103
Title: BiVACOR® Total Artificial Heart Early Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BiVACOR Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CP-0001
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure; Biventricular Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- BiVACOR TAH (Experimental): The BiVACOR TAH System will be implanted as a bridge to transplant (BTT) for adults with severe irreversible biventricular heart failure or univentricular heart failure in which LVAD support is not recommended, and who are eligible for cardiac transplantation.
  Interventions: Device: BiVACOR TAH System

INTERVENTIONS:
Device: BiVACOR TAH System — The BiVACOR pump is an implantable rotary biventricular blood pump that uses magnetic levitation technology for increased durability to replace both ventricles of a failing heart. The device is intended to replace the diseased heart in patients suffering from heart failure to bridge the time to heart transplant.

SUMMARY:
The purpose of this study is to assess the feasibility of using the BiVACOR Total Artificial Heart (TAH) System to support adult patients with severe biventricular heart failure, or univentricular heart failure in which left ventricular assist device (LVAD) support is not recommended, who require mechanical circulatory support to sustain life. The BiVACOR TAH System is intended for use as a bridge to transplant (BTT). Feasibility will be assessed by evaluating safety and performance of the BiVACOR TAH System in study subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patient has severe, irreversible biventricular heart failure and is eligible for biventricular mechanical circulatory support based on the International Society of Heart and Lung Transplantation (ISHLT) guidelines or has univentricular heart failure in which LVAD support is not recommended. ISHLT Guidelines for Biventricular Support:

  1. Biventricular failure with at least two of the following hemodynamic and/or echocardiographic measurements.

     1. Right ventricular ejection fraction (RVEF) ≤ 30%
     2. Right ventricular stroke work index (RVSWI) ≤ 0.25 g/m/beat/m2
     3. Tricuspid annular plane systolic excursion (TAPSE) ≤ 14 mm
     4. Right ventricular (RV) to left ventricular (LV) end-diastolic diameter ratio > 0.72
     5. Central venous pressure (CVP) > 15mmHg
     6. CVP to pulmonary capillary wedge pressure (PCWP) ratio > 0.63
     7. Tricuspid insufficiency grade 4
     8. Pulmonary artery pressure index (PAPi) < 2
  2. Treatment-refractory recurrent and sustained ventricular tachycardia or ventricular fibrillation in the presence of untreatable arrhythmogenic pathologic substrate.
  3. Heart failure due to restrictive or constrictive physiology (e.g., hypertrophic cardiomyopathy, cardiac amyloidosis/senile or other infiltrative heart disease).
* Patient is categorized as INTERMACS Patient Profile Classification 2 or 3.
* Patient is classified as NYHA Class IV.
* Patient has a left ventricular ejection fraction (LVEF) ≤ 25%, with the exception of patients with restrictive or constrictive physiology.
* Patient is inotrope dependent, OR has a cardiac index (CI) ≤ 2.2 L/min/m2 without inotropes if inotropes are contraindicated (e.g., restrictive or constrictive heart failure), and meets one of the following criteria:

  1. Is on optimal medical management (OMM), based on current heart failure practice guidelines for at least 45 out of the last 60 days and is failing to respond or is not able to tolerate OMM; or
  2. Has advanced heart failure for at least 14 days and is dependent on an intra-aortic balloon pump (IABP) or similar temporary mechanical circulatory support device (MCSD) for at least seven days.
* Patient is eligible for cardiac transplantation as determined by the implanting center.
* Patient has adequate room in the chest as determined by 3-D imaging or other standard clinical assessments.
* Patient has read and understands the informed consent form (ICF) and has voluntarily provided informed consent.

Exclusion Criteria:

* Patient has contraindications to anticoagulation or antiplatelet therapies.
* Patient has coagulopathy defined by a platelet count < 50 k/µl.
* Patient has insufficient space in the chest to accommodate the BiVACOR pump.
* Patient has a body mass index (BMI) ≥ 35 kg/m2.
* Patient is highly pre-sensitized prior to pump implantation.
* Patient is unconscious and unresponsive.
* Patient is on pre-implant extracorporeal membrane oxygenation (ECMO) for > 7 days.
* Patient is on pre-implant temporary MCSD for more than 21 days [e.g., Intra-aortic balloon pump (IABP), Impella, CentriMag, etc.] unless ambulatory and free from adverse effects associated with the MCSD.
* Patient is implanted with durable mechanical circulatory support (LVAD or RVAD).
* Patient experienced cerebrovascular accident (CVA) within three months of eligibility evaluation.
* Patient has severe end-organ dysfunction as evidenced by:

  1. Total bilirubin > 4.0 mg/dL or cirrhosis confirmed by imaging or positive biopsy, and/or
  2. Glomerular filtration rate (GFR) < 30 mL/min/1.73 m2 or renal replacement therapy dependence.
* Patient has severe chronic obstructive pulmonary disease (COPD) or restrictive lung disease requiring home oxygen.
* Patient has primary pulmonary hypertension ≥ 8 Wood units.
* Patient has severe systemic light-chain amyloidosis.
* Patient has been diagnosed with severe cardiac cachexia or irreversible frailty.
* Patient has diabetes with advanced diabetic neuropathy with accompanying skin ulceration.
* Patient has a blood-borne infection within seven days of eligibility evaluation. Positive blood cultures reflective of contaminants (e.g., Staphylococcus epidermidis) will not be considered an exclusion.
* Patient is pregnant or planning pregnancy.
* Patient has a co-morbidity or illness that would limit survival to less than two years.
* Patient has a current drug and/or alcohol addiction or known substance abuse.
* Patient has insufficient social support or a history of non-compliance with medical instructions as determined by the Investigator.
* Patient is participating in another clinical trial that may impact or confound the results of the BiVACOR TAH EFS.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility Endpoint | 6 months or time of heart transplant (if prior to 6 months post pump implant)
  Survival on the original BiVACOR pump
Safety Endpoint | Through 6 months
  Evaluation of the safety of the BiVACOR TAH System using INTERMACS adverse event (AE) terms and definitions (INTERMACS Manual of Operations Version 5).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Banner - University Medical Center Phoenix, Phoenix, Arizona
  - Duke University Hospital, Durham, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Texas Heart Institute / Baylor St. Luke's Medical Center, Houston, Texas